CLINICAL TRIAL: NCT05770089
Title: Impact of an Adapted Physical Activity Program Supervised by Videoconference in Patients With Anorexia Nervosa: a Pilot Study
Brief Title: Videoconferencing Adapted Physical Activity in Anorexia Nervosa: a Pilot Study
Acronym: APAREXIM-P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A01245-38
Record Dates: First submitted 2022-12-13; First posted 2023-03-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa; Exercise Therapy; Videoconferencing
Keywords: eating disorders; anorexia nervosa; physical activity; exercise; psychiatry; mental health; muscle strength; chronobiology; physical condition; adolescent; pediatric; videoconferencing
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AM-APA (Experimental): The group following the Adapted Physical Activity program via videoconferencing in addition to the outpatient care.
  Interventions: Other: Adapted Physical Activity (APA)
- AM-T (No Intervention): The group without additional intervention other than the outpatient care.

INTERVENTIONS:
Other: Adapted Physical Activity (APA) — A 8-weeks program of APA (2x1hour per week) via videoconferencing composed of resistance training and yoga.
  Other Names: Interventional exercise therapy
  Arms: AM-APA

SUMMARY:
The primary objectives of the APAREXIM'Pilot study are to evaluate the short- and medium-term effects of a live supervised Adapted Physical Activity (APA) program via videoconferencing on:

* Feasibility and acceptability of APA via videoconferencing by the patients.
* The primary symptoms of Anorexia Nervosa (AN).

The secondary objectives are to evaluate the impact of this program on :

* Mental health
* Physical condition
* Sleep-wake cycle (sleep disturbance and physical hyperactivity)

The patients will first undergo an inclusion visit (T0) at the University Hospital of Caen, then a first evaluation session (T1) at the COMETE laboratory in Caen (physical tests, questionnaires, sleep diary, actimetry). They will then be randomly divided into 2 groups: 15 patients who will follow an APA program supervised by videoconference for 8 weeks (AM-APA) at their home, in addition to the usual outpatient treatment, and 15 patients who will benefit only from the classic outpatient treatment (AM-T). All patients will undergo two additional evaluation sessions at one week post-program (T2) and at 3 months post-program (T3).

DETAILED DESCRIPTION:
Background: Anorexia nervosa (AN) is an eating disorder (ED), mainly in women, characterized by strict and voluntary food deprivation over a long period of time, which can last from several months to several years, leading to significant weight loss. This disease affects 2.2 to 4% of the general population in Europe and is one of the most fatal psychiatric diseases in people under 25 years old. Physiological and psychological disorders are very often associated with AN, as well as an alteration of the sleep-wake cycle. In order to reduce the risk of chronicity of the disease and to prevent its various complications in young women, early and multidisciplinary therapeutic management is recommended by public health authorities. However, this management remains long and complex due to the diversity and severity of the symptoms, a lack of adherence of patients to treatment protocols, but also a lack of therapeutic continuity after hospitalization. Recently, new non-medicinal therapies based on Adapted Physical Activity (APA) have been developed to prevent and reduce the main symptoms of AN and associated disorders in an effective and lasting way. However, to our knowledge, interventional research in this field remains scarce and presents limited results. Furthermore, the scientific literature does not report any evaluation of the feasibility, acceptability, and effectiveness of a home video-conference-supervised APA intervention with AN patients.

Objectives: The primary objectives of the APAREXIM'Pilot study are to evaluate the short- and medium-term effects of a live supervised APA program via videoconferencing on feasibility and acceptability of APA via videoconferencing by the patients and the primary symptoms of AN. The secondary objectives are to evaluate the impact of this program on mental health, physical condition and the sleep-wake cycle (sleep disturbance and physical hyperactivity), as well as its.

Method: This randomized controlled intervention study will be conducted with 30 adolescent and young adult girls with AN. The patients will first undergo an inclusion visit (T0) at the University Hospital of Caen, then a first evaluation session (T1) at the COMETE laboratory in Caen (physical tests, questionnaires, sleep diary, actimetry). They will then be randomly divided into 2 groups: 15 patients who will follow an APA program supervised by videoconference for 8 weeks (AM-APA) at their home, in addition to the usual outpatient treatment, and 15 patients who will benefit only from the classic outpatient treatment (AM-T). All patients will undergo two additional evaluation sessions at one week post-program (T2) and at 3 months post-program (T3).

Perspectives: The results obtained will allow to evaluate the acceptability and the feasibility of a distance APA program, and to bring additional evidence of the effectiveness of an APA intervention in patients with AM, as well as elements of understanding of the regulation of this pathology by APA. In addition, the APAREXIM'Pilot study will allow to test and validate an APA program for patients with AM, which could eventually be integrated in the management of patients on the national territory.

ELIGIBILITY:
Inclusion Criteria:

* Female patient between 13 and 18 years old, with typical anorexia nervosa symptoms diagnosed by a specialist.
* Patient followed in outpatient care.
* Collection of the signature of the informed consent.
* Patient affiliated to the health insurance system.
* Agreement of the legal representatives

Exclusion Criteria:

* Patient with contraindications to physical activity or with a state of health judged critical by the doctor.
* Person deprived of liberty by judicial or administrative decision, or under guardianship or curatorship.
* Pregnant or breast-feeding woman.
* Patient included in another biomedical research protocol during the present study.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability and Preferences questionnaire (TAP-Q) | T2 (just after the APA program)
  Questionnaire (scale) assessing the acceptability of the APA program via videoconferencing (high score mean better outcome).
Eating Attitude Test - 26 (EAT-26) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing the severity of main anorexic symptoms (high score mean worse outcome).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression (HAD) scale | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing anxious and depressive symptoms (high score mean worse outcome).
Rosenberg Self-esteem Scale (RSS) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing self-esteem (high score mean better outcome).
Contour Drawing Rating Scale (CDRS) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing self-esteem (high score mean worse outcome).
Body Esteem Scale (BES) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing body esteem (high score mean better outcome).
Exercise Dependence Scale Revised | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing exercise dependence (high score mean worse outcome).
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing interoceptive awareness (high score mean better outcome).
Pittsburgh Sleep Quality Index (PSQI) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Questionnaire (scale) assessing sleep quality (high score mean worse outcome).
Actimetry | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  One week of actimetry with an accelerometer watch measuring 7x24h activity counts allowing to extract day and night activity level.
Body Mass Index (BMI) | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Measure of body weight and height to compute the BMI
Body composition - Body cellular mass | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Bio-impedance measuring of body cellular mass
Body composition - Fat mass | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Bio-impedance measuring of body fat mass
Body composition - Fat free mass | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Bio-impedance measuring of body fat-free mass
Body composition - Total body water | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Bio-impedance measuring of total body water
Body composition - Extracellular water | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Bio-impedance measuring of body extracellular water
Isokinetic assessment of upper and lower limbs | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Isokinetic peak torque (concentric contraction at 60°/sec and 240°/sec) of forearm and leg flexion/extension.
Back extension strength | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Assessment of the back extension strength with a dynamometer
Shirado test | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Assessment of the isometric back flexion endurance with the Shirado test
Sorensen test | Change from T1 (just before the APA program) at T2 (just after the APA program) then T3 (8 weeks after the APA program)
  Assessment of the isometric back extension endurance with the Sorensen test

CONTACTS AND LOCATIONS:
Overall Officials: Fabian GUENOLE, MD PhD Pr, Principal Investigator — Caen Hospital University
Locations (1):
- Caen University Hospital, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No